CLINICAL TRIAL: NCT02924142
Title: Treatment Outcomes Based on Patient's Oral Health Related Quality of Life (OHRQoL) After Receiving Conventional Clasp or Precision Attachment Removable Partial Dentures in Distal Extension Cases: A Randomized Controlled Clinical Trial
Brief Title: Treatment Outcomes After Receiving Conventional Clasp or Precision Attachment Removable Partial Dentures.
Acronym: OTCap
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rania Hassan, Dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2016-09-212
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Bilateral Edentulous Mandible (Kennedy Class I)
Keywords: Kennedy classification for edentulous ridge

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Mandibular removable partial denture with OT Cap attachment
  Interventions: Device: OT Cap attachment
- Comparator (No Intervention): Mandibular removable partial denture with gingival approaching clasp assembly

INTERVENTIONS:
Device: OT Cap attachment — The RHEIN 83 OT CAP attachment system is an extra-coronal castable attachment positioned on the distal of the abutment crowns as an extension allowing a lot of vertical space for optimal esthetics.
  Arms: Intervention

SUMMARY:
PICOTS:

P: Kennedy class І patients

I : Mandibular removable partial denture with OT Cap attachment

C: Mandibular removable partial denture with gingival approaching clasp assembly

O: 1ry outcome: Oral Health Related Quality of Life

2ry outcome: Biting force

T: 1 Year

S : Randomized control trial

Research question:

In Kennedy class І patients will the removable partial denture with OT Cap attachment compared to conventional removable partial denture with clasp assembly results in difference in Oral Health Related Quality of Life of Patients?

DETAILED DESCRIPTION:
In bilateral edentulous mandible with missing molars, the clasp retained partial denture will be compared with precision attachment partial denture for better quality of life for patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with mandibular free end saddle cases.
2. Patients less than 75 years old.
3. Patients who approved to be included in the trial and signed the informed consent.
4. Patients are not suffering from diabetes mellitus.

Exclusion Criteria:

1. Patients are suffering from diabetes mellitus.
2. Patients above 75 years old.
3. Patients are receiving chemotherapy or radiotherapy.
4. Patients with severe Temporomandibular Joint problems.
5. Patients who refused the trial.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Oral Health Related Quality of Life | 1 Year
  Questionnaire

SECONDARY OUTCOMES:
Biting force | 1 Year
  i-load Star Sensor

CONTACTS AND LOCATIONS:
Overall Officials: Yousr M. Mady, Professor, Study Director — Faculty of Oral and Dental Medicine, Cairo University, Cairo, Egypt; Ahmed M. Fayyad, A. Professor, Study Director — Faculty of Oral and Dental Medicine, Cairo University, Cairo, Egypt
Locations (1):
- Faculty of Oral and Dental Medicine, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided